CLINICAL TRIAL: NCT07392788
Title: Early Gliflozin Treatment in Elderly Patient Hospitalized for Decompensated Chronic Heart Failure Admitted in the Emergency Room - a Feasibility Study
Brief Title: Early Gliflozin for Elderly Patients With Acute Decompensated Heart Failure in the Emergency Department
Acronym: GlifloFastER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024/882
Record Dates: First submitted 2024-11-14; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Acute Heart Failure (AHF)
Keywords: acute heart failure; emergency department; elderly; SGLT2 Inhibitors; Feasibility study; Acute Decompensated Chronic Heart Failure
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): * Early initiation of dapagliflozin 10mg daily within 24h of ED admission
  * Telephone follow-up by cardiac nurse practitioner at 1 month
  * Standard acute decompensated heart failure care
  Interventions: Drug: Early initiation of dapagliflozin 10mg daily within 24h of emergency department admission; Other: Telephone follow-up by cardiac nurse practitioner at 1 month; Other: Standard acute decompensated heart failure care
- Control group (Active Comparator): ✓ Standard acute decompensated heart failure care ONLY
  Interventions: Other: Standard acute decompensated heart failure care

INTERVENTIONS:
Drug: Early initiation of dapagliflozin 10mg daily within 24h of emergency department admission — Early initiation of dapagliflozin 10mg daily within 24h of ED admission
  Arms: Intervention group
Other: Telephone follow-up by cardiac nurse practitioner at 1 month — Telephone follow-up by cardiac nurse practitioner at 1 month
  Arms: Intervention group
Other: Standard acute decompensated heart failure care — Standard acute decompensated heart failure care

SUMMARY:
Background: SGLT2 inhibitors reduce CHF morbidity/mortality but are underutilized in elderly patients with acute decompensated CHF (ADCHF) admitted outside cardiology departments.

Objective: Assess feasibility of early ED-initiated gliflozin therapy in elderly ADCHF patients.

Design: Multicenter, randomized, open-label pilot study; N=144 patients (72 per arm) across 6 EDs over 30 months.

Population: Age ≥75 years, ED admission for ADCHF (symptomatic worsening, congestion, elevated natriuretic peptides), gliflozin-naïve, requiring hospitalization.

Key Exclusions: Type 1 diabetes, eGFR <25 mL/min/1.73m², cardiogenic shock, recent ACS, cardiology ward admission.

Intervention:

Treatment: Dapagliflozin 10mg daily within 24h + cardiac nurse telephone follow-up at 1 month Control: Standard care only Primary Outcome: Feasibility (organizational implementation, acceptability, protocol adherence, timeline compliance).

Follow-up: 7-day visit (clinical assessment, NT-proBNP, echocardiography) and 3-month cardiology consultation (mortality, rehospitalization, QoL, biomarkers, safety parameters).

DETAILED DESCRIPTION:
Rationale: Chronic heart failure (CHF) in elderly patients is associated with increased mortality, rehospitalization risk, and significant quality of life impairment. SGLT2 inhibitors (gliflozins) have demonstrated efficacy in reducing morbidity and mortality in stabilized CHF patients when initiated 24-72 hours after emergency department (ED) admission in cardiology units. However, most elderly CHF patients presenting to the ED with acute decompensation are hospitalized in non-cardiology departments and do not receive optimal therapeutic management including gliflozins, despite their potential significant benefit in this population.

Hypothesis: Early initiation of gliflozins in the ED setting, without waiting for cardiology consultation, could avoid potential delays in optimal treatment for elderly patients with acute decompensated chronic heart failure (ADCHF).

Study Design: This is a multicenter, prospective, randomized, open-label, parallel-group feasibility pilot study conducted over 30 months (including 12 months of recruitment) across 6 hospital emergency departments in France. The study will evaluate the overall feasibility of early ED initiation of gliflozins plus telephone follow-up compared to standard care in elderly patients admitted for ADCHF who are not previously treated with gliflozins.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 75 years
2. ED admission for ADCHF with:

   * Worsening CHF symptoms (dyspnea, fatigue, weight gain, edema)
   * Objective signs of peripheral/pulmonary congestion
   * Elevated natriuretic peptides:

     * Sinus rhythm: BNP ≥ 400 pg/mL or NT-proBNP ≥ 1,600 pg/mL
     * Atrial fibrillation: BNP ≥ 600 pg/mL or NT-proBNP ≥ 2,400 pg/mL
   * Need for treatment intensification
3. Expected hospitalization
4. No prior gliflozin treatment
5. Signed informed consent

Exclusion Criteria:

* Type 1 diabetes
* Chronic kidney disease (eGFR < 25ml/min/1.73m²)
* Cardiogenic shock
* Acute coronary syndrome (current or within 30 days)
* Severe valvular disease requiring surgery
* Recent/planned coronary intervention
* Known intolerance to study medication
* Legal protection measure or inability to consent
* Hospitalization in cardiology department
* Discharge home or to nursing home

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Organizational feasibility: Implementation of procedures | 3 months
  Successful implementation of study procedures (yes/no). Binary assessment of whether study procedures were successfully implemented at each site.
Organizational feasibility: Patient flow assessment | 3 months
  Proportion of eligible patients successfully enrolled. Ratio of patients enrolled to patients screened, expressed as percentage.
Acceptability: Number of refusals | 3 months
  Number of patients refusing participation. Total count of eligible patients who declined to participate.
Acceptability: Reasons for refusal | 3 months
  Categories of refusal reasons. Qualitative categorization of stated reasons for study refusal.
Protocol adherence: Attrition rate | 3 months
  Proportion of participants completing the study protocol. Percentage of enrolled patients who complete all protocol requirements without withdrawal.
Protocol adherence: CRF completion rate | 3 months
  Case report form completion rate. Percentage of required case report form fields completed across all participants.
Protocol adherence: Telephone follow-up success rate | 1 month
  Proportion of patients successfully contacted by telephone at 1 month. Percentage of intervention group patients successfully reached for telephone follow-up by cardiac nurse practitioner.
Timeline adherence | 3 months
  Study timeline compliance (yes/no). Binary assessment of whether study met anticipated timeline for recruitment and follow-up phases.

CONTACTS AND LOCATIONS:
Overall Officials: Fatimata SARR, PhD, Study Chair — CHU Besançon; Frédéric MAUNY, MD, PhD, Study Chair — CHU Besançon; Marc PUYRAVEAU, MSc, Study Chair — CHU Besançon; Thibaut DESMETTRE, MD, PhD, Study Chair — University Hospital, Geneva; Johan COSSUS, MD, Study Chair — CHU Besançon

IPD SHARING:
Plan to Share IPD: Yes
Plan Description:
  De-identified individual participant data (IPD) that underlie the results reported in published articles, including the study protocol, statistical analysis plan, and informed consent form, may be shared upon reasonable request after study completion and primary publication.
  Access Criteria:
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After study completion and primary publication.
Access Criteria: IPD may be available to researchers who provide a methodologically sound proposal for academic purposes. Requests should be directed to [principal investigator email]. Requestors will need to sign a data access agreement and obtain approval from their local ethics committee. Data will be shared in compliance with EU GDPR and French data protection regulations.